CLINICAL TRIAL: NCT00014183
Title: A Phase II Study Of ZD1839 (NSC #715055) In Renal Cell Carcinoma Stage IV And Renal Cell Carcinoma Recurrent
Brief Title: ZD 1839 in Treating Patients With Stage IV or Recurrent Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068512; MSGCC-0044; NCI-1639
Record Dates: First submitted 2001-04-10; First posted 2004-01-01 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as ZD 1839 may interfere with the growth of the tumor cells and slow the growth of kidney cancer.

PURPOSE: Phase II trial to study the effectiveness of ZD 1839 in treating patients who have recurrent or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with progressive stage IV or recurrent renal cell cancer treated with ZD 1839.
* Determine the median time to objective progression in these patients receiving this drug.
* Determine the toxic effects of this drug in this patient population.
* Determine if epidermal growth factor receptor expression in tumor tissue correlates with response and survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive oral ZD 1839 daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 21-45 patients will be accrued for this study within 11-23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV or recurrent renal cell carcinoma not amenable to potentially curative surgery
* Evidence of disease progression
* Measurable disease

  * At least 20 mm with conventional techniques OR
  * At least 10 mm with spiral CT scan
* No brain metastases
* Malignant tissue available

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No prior allergy to compounds of similar chemical or biologic composition to ZD 1839
* No ongoing or active infection
* No other uncontrolled illness or psychiatric condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 2 prior immunotherapy (interferon alfa or interleukin-2) regimens
* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunotherapy

Chemotherapy:

* No more than 1 prior chemotherapy regimen
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No prior therapy for metastatic disease
* No other concurrent investigational agents
* No concurrent oral retinoids

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2002-05 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Dawson, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland